CLINICAL TRIAL: NCT01150851
Title: Oxidative Stress in Chronic Kidney Disease: Diet and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 100716
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- caloric restriction (Active Comparator): 10 to 15% reduction in total daily calories (300 to 500 kcal reduction) from the usual daily energy consumption for 4 months duration
  Interventions: Other: caloric restriction
- aerobic exercise (Active Comparator): supervised physical activity for a maximum of 30-45 minutes, 3 times per week for 4 months duration
  Interventions: Other: aerobic exercise
- caloric restriction and aerobic exercise (Active Comparator): 10 to 15% reduction in total daily calories (300 to 500 kcal reduction) from the usual daily energy consumption for 4 months duration, and supervised physical activity for a maximum of 30-45 minutes, 3 times per week for 4 months duration
  Interventions: Other: caloric restriction; Other: aerobic exercise
- usual diet and usual activity (No Intervention): usual diet and usual activity

INTERVENTIONS:
Other: caloric restriction — 10 to 15% reduction in total daily calories (300 to 500 kcal reduction) from the usual daily energy consumption for 4 months duration
  Arms: caloric restriction; caloric restriction and aerobic exercise
Other: aerobic exercise — supervised physical activity for a maximum of 30-45 minutes, 3 times per week for 4 months duration
  Arms: aerobic exercise; caloric restriction and aerobic exercise

SUMMARY:
The central aim of this study is to improve understanding of how metabolic pathways that contribute to adiposity also amplify risks of kidney disease progression and cardiovascular disease in subjects with moderate to severe CKD. In order to achieve this goal, we propose the following aims through a randomized 2x2 factorial design trial in subjects with moderate to severe CKD: (a) To assess the feasibility of implementing aerobic exercise and caloric restriction interventions, and (b) To examine the effects of aerobic exercise and caloric restriction on a metabolic risk profile, including systemic measures of oxidative stress, inflammation, insulin resistance, and endothelial dysfunction.

Hypothesis: We hypothesize that implementation of caloric restriction and aerobic exercise is feasible and can improve the metabolic milieu (as assessed by measures of oxidative stress, inflammation, insulin resistance, and endothelial dysfunction) in subjects with moderate to severe CKD.

Interim analysis may be performed (no specific plan at this time).

ELIGIBILITY:
Inclusion Criteria:

* Stage III-IV CKD measured by the MDRD equation with eGFR 15-60 ml/min/1.73m2;
* Age 18-75 years;
* BMI ≥ 25;
* Life expectancy ≥ 1 year;
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Any acute inflammatory condition (including chronic infection requiring treatment, and collagen vascular disease including active gout);
* Pregnancy;
* Taking high-dose anti-oxidants (Vitamin E or C);
* Chronic use of anti-inflammatory medication except low dose (< 10mg/d) prednisone and aspirin (< 100 mg/day);
* Significant cardiac or vascular disease (symptomatic disease or CV event including congestive heart failure within 6 months);
* Significant occlusive atherosclerotic disease or ischemic disease (on non-invasive or invasive diagnostic procedures);
* Significant physical immobility or disabilities (joint replacement, muscular disorders);
* Type I diabetes mellitus, or Type II requiring insulin therapy;
* History of poor adherence to medical regimen;
* Those subjects who have a diagnosis of atrial fibrillation or a pacemaker will be allowed in the study but will not undergo Arterial Tonometry (PWV) studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
a change in plasma F-2-isoprostane concentration | baseline and 4 months
a change in VO2 max | baseline and 4 months
a change in weight | baseline and 4 months
a change in absolute fat mass | baseline and 4 months

SECONDARY OUTCOMES:
a change in biomarkers of inflammation | baseline and 4 months
a change in biomarkers of endothelial dysfunction | baseline and 4 months
a change in biomarkers of insulin resistance | baseline and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University; Jonathan Himmelfarb, MD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Springfield College, Springfield, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kidney Research Institute, Seattle, Washington
  - Providence Sacred Heart Medical Research Center, Spokane, Washington

REFERENCES:
- [Derived] Jaramillo-Morales J, Korucu B, Pike MM, Lipworth L, Stewart T, Headley SAE, Germain M, Begue G, Roshanravan B, Tuttle KR, Himmelfarb J, Robinson-Cohen C, Ikizler TA, Gamboa JL. Effects of caloric restriction and aerobic exercise on circulating cell-free mitochondrial DNA in patients with moderate to severe chronic kidney disease. Am J Physiol Renal Physiol. 2022 Jan 1;322(1):F68-F75. doi: 10.1152/ajprenal.00270.2021. Epub 2021 Nov 29. PMID 34843657
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Aydemir N, Pike MM, Alsouqi A, Headley SAE, Tuttle K, Evans EE, Milch CM, Moody KA, Germain M, Lipworth L, Himmelfarb J, Ikizler TA, Robinson-Cohen C. Effects of diet and exercise on adipocytokine levels in patients with moderate to severe chronic kidney disease. Nutr Metab Cardiovasc Dis. 2020 Jul 24;30(8):1375-1381. doi: 10.1016/j.numecd.2020.04.012. Epub 2020 Apr 21. PMID 32571614